CLINICAL TRIAL: NCT06119828
Title: THE EFFECT OF BREASTFEEDING EDUCATıON ON BREASTFEEDING PARAMETERS GIVEN TO FAMILY MEMBERS PROVIDING SUPPORT TO THE MOTHER IN THE POSTPARTUM PERİOD
Brief Title: The Effect of Breastfeeding Education Given to Family Members on Breastfeeding Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Cevriye Ocaktan Tetikçok, Research assistant, Selcuk University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019/706
Record Dates: First submitted 2023-10-27; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Breastfeeding
Keywords: family member, breastfeeding self-efficacy, nutritional attitude
MeSH Terms: conditions — Breast Feeding | interventions — Educational Status; Control Groups

STUDY DESIGN:
Intervention Model Description: It was conducted as a randomized controlled experimental study to determine the effect of breastfeeding education given to the family member who supports the mother in the postpartum period on breastfeeding parameters.
Masking Description: Since one researcher conducted the study, blinding was not possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parallel Asignment (Experimental): Power analysis was performed using the G*Power(v3.1.9) program to determine the sample size. The power of the study is expressed as 1-β (β = probability of type II error) and in general, studies must have 80% power. According to the effect size coefficients determined by Cohen, assuming that the evaluations to be made between two independent groups will have a medium effect size (d = 0.5), α = 0.05 and β = 0.20, it was determined that there should be at least 64 people in each group, according to the calculation.
  Interventions: Behavioral: breastfeeding education for family members; Other: receiving routine breastfeeding training

INTERVENTIONS:
Behavioral: breastfeeding education for family members — The first breastfeeding skills of mothers who gave birth in the delivery room and the first breastfeeding skills after birth were evaluated using BEDÖ. After giving birth, mothers were taken to the maternity ward after being kept under control in the delivery room for 2 hours. After the mothers' 1-hour breastfeeding was evaluated in the delivery room, the training phase of family members began. CBT was administered to family members in the waiting room before the training, which lasted approximately 7-8 minutes. Then, breastfeeding training was given to family members for 20-25 minutes. BBST was applied after the mother transferred to the maternity ward. Before the mother and the baby were discharged from the hospital, BEDÖ and BBTÖ were administered to the family member. On the 15th postpartum day, the family member was called by phone and reminded about breastfeeding education. At the first month postpartum,Checklist were administered to the mother via telephone conversation
  Other Names: education
Other: receiving routine breastfeeding training — After giving birth, mothers were taken to the maternity ward after being kept under control in the delivery room for 2 hours. Mothers' breastfeeding was evaluated at the 1st hour in the delivery room. CBT was administered to family members in the waiting room. BBST was applied after the mother transferred to the maternity ward. Before the mother and the baby were discharged from the hospital, BEDÖ and BBTÖ were administered to the family member. At the first month postpartum, BBTÖ was administered to the family member, and BBTÖ and EÖY scale and Breastfeeding Checklist were administered to the mother over the phone.
  Other Names: Control groups

SUMMARY:
The Effect of Breastfeeding Education Given to Family Members Who Support the Mother in the Postpartum Period on Breastfeeding Parameters. Istanbul University-Cerrahpaşa Graduate Education Institute, Midwifery Department. Doctoral Thesis. Istanbul.

I To examine the effect of breastfeeding education given to family members in the postpartum period on breastfeeding parameters. It was conducted as a randomized controlled experimental study to determine the effect of breastfeeding education given to the family member who supports the mother in the postpartum period on breastfeeding parameters

DETAILED DESCRIPTION:
Power analysis was performed using the G*Power(v3.1.9) program to determine the sample size. The power of the study is expressed as 1-β (β = probability of type II error) and in general, studies must have 80% power. According to the effect size coefficients determined by Cohen, assuming that the evaluations to be made between two independent groups will have a medium effect size (d = 0.5), α = 0.05 and β = 0.20, it was determined that there should be at least 64 people in each group, according to the calculation. Considering that there may be losses during the study process, the sample size was increased by 20% and it was decided to include at least 77 people in each group. The calculation of the sample size was based on Zeliha Burcu Baysal's doctoral thesis titled The Effect of Breastfeeding Education and Counseling Given to Pregnant Women and Their Spouses on the Breastfeeding Process and Attachment.

The main aims of the study are:

Breastfeeding education given to the family member; Does it increase the rate of mothers starting breastfeeding? Breastfeeding education given to the family member; Does it increase the rate of mothers giving exclusive breastfeeding in the first month? In the intervention group, family members will be given breastfeeding education and they will be asked to support mothers in the postpartum period.

In the comparison group, no breastfeeding education was given to the family member.

ELIGIBILITY:
Inclusion Criteria:

For mothers;

* Will receive support from a family member during the postpartum period,
* Having an uncomplicated pregnancy and birth history,
* No multiple pregnancy,
* Not giving birth before the 37th week of pregnancy,
* Not having any disease that prevents breastfeeding in the postpartum period (undergoing chemotherapy, active tuberculosis, using drugs that prevent breastfeeding, etc.),
* Spending the pregnancy period and the first month after birth in the area where the research will be conducted,
* Being at least a primary school graduate,
* No communication problems,
* Being primiparous or multiparous with breastfeeding problems,
* For the family member who will provide support to the mother in the postpartum period, as long as the baby does not have any health problems that prevent breastfeeding;
* Spending time with the mother regularly for at least 1 hour at least five days a week during the postpartum period,
* Being able to communicate in Turkish,
* It was defined as residing in the same city during the period when the research data was collected.

Exclusion Criteria:

For mothers;

* Those with a history of complicated pregnancy and birth,
* Those with multiple pregnancies,
* Those with premature babies,
* Conditions related to mother and baby that prevent breastfeeding in the postpartum period (pregnancy psychosis, congenital anomaly, sucking and swallowing coordination disorder, etc.),
* Those who will not live in the area where the research will be conducted during pregnancy and the first month after birth,
* Those who have difficulty communicating for various reasons (not being able to speak Turkish, serious hearing problems, etc.)
* Mothers who did not meet the research criteria for any reason after being included in the study (interventional birth, the baby having any disease requiring hospitalization in neonatal intensive care, etc.) were excluded from the scope of the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
breastfeeding education given to family members | postpartum 1st month
  Breastfeeding education given to the family member; Does it increase the rate of mothers starting breastfeeding? Breastfeeding education given to the family member; Does it increase the rate of mothers giving exclusive breastfeeding in the first month?

CONTACTS AND LOCATIONS:
Locations (1):
- SelcukUniversity, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There are no plans for use by other workers.

REFERENCES:
- [Result] Holbrook KE, White MC, Heyman MB, Wojcicki JM. Maternal sociodemographic characteristics and the use of the Iowa Infant Attitude Feeding Scale to describe breastfeeding initiation and duration in a population of urban, Latina mothers: a prospective cohort study. Int Breastfeed J. 2013 Jul 8;8(1):7. doi: 10.1186/1746-4358-8-7. PMID 23835065
- [Result] Han FL, Ho YJ, McGrath JM. The influence of breastfeeding attitudes on breastfeeding behavior of postpartum women and their spouses. Heliyon. 2023 Feb 23;9(3):e13987. doi: 10.1016/j.heliyon.2023.e13987. eCollection 2023 Mar. PMID 36879970
- [Result] Houghtaling B, Byker Shanks C, Ahmed S, Rink E. Grandmother and health care professional breastfeeding perspectives provide opportunities for health promotion in an American Indian community. Soc Sci Med. 2018 Jul;208:80-88. doi: 10.1016/j.socscimed.2018.05.017. Epub 2018 May 8. PMID 29772397